CLINICAL TRIAL: NCT01206569
Title: Long-Acting Tacrolimus for the Treatment of Resistant Lupus Nephritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFKLN
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Lupus Nephritis
Keywords: glomerulonephritis; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Nephritis; Glomerulonephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- advagraf (Experimental): Long-acting tacrolimus (Advagraf, Astellas Pharma) will be started at single daily dose of 0.15-0.2 mg/kg/day for 6 months.
  Interventions: Drug: Long-acting tacrolimus (Advagraf, Astellas Pharma)

INTERVENTIONS:
Drug: Long-acting tacrolimus (Advagraf, Astellas Pharma) — Long-acting tacrolimus (Advagraf, Astellas Pharma) will be started at single daily dose of 0.15-0.2 mg/kg/day for 6 months.

SUMMARY:
Glomerulonephritis is one of the major disease manifestations of systemic lupus erythematosus (SLE). Around one-third of the patients, however, do not respond to conventional immunosuppressive therapy, and they have a high risk of progressing to dialysis-dependent renal failure. Recent studies suggest that immunosuppressive therapy targeted against the calcineurin pathway of T-helper cell, for example, tacrolimus, may be effective in the treatment of primary glomerulonephritis. The investigators plan to an open-label single-arm study the efficacy and safety of long-acting tacrolimus in the treatment of treatment-resistant lupus nephritis. Twenty-five patients with biopsy-proven lupus nephritis will be recruited. They will be treated with oral prednisolone and long-acting tacrolimus for 6 months, followed by 6 months of maintenance steroid and azathioprine. Proteinuria, renal function, clinical and serologic lupus activity will be monitored. This study will explore the potential role of long-acting tacrolimus in resistant lupus nephritis, which has a poor prognosis and no effective treatment at the moment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 with informed consent.
* Fulfill the revised American College of Rheumatology criteria for SLE
* Biopsy-proven class III, IV, or V lupus nephritis within the past 24 months.
* Could not achieve complete remission after at least 4 months of conventional therapy (oral steroid plus cyclosphosphamide or mycophenolate mofetil).
* NB. Complete response is defined as proteinuria less than 0.5 g/day, with normal urinary sediment, a normal serum albumin concentration, and serum creatinine <15% above the base-line value.
* Female patients of child-bearing age and male patients agree to maintain effective birth control practice during the study.

Exclusion Criteria:

* Abnormal liver function tests
* Hepatitis B surface antigen or hepatitis C antibody positive
* Diabetic
* Receiving NSAID or other agents known to influence urinary
* Protein excretion
* Allergic or intolerant to macrolide antibiotics or tacrolimus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
overall clinical response | 6 months
  complete response is defined as urinary protein < 0.5 g/day, with normal urinary sediment, normal serum albumin, and serum creatinine < 15% above the base-line value. Partial response is defined as urinary protein between 0.6 and 2.9 g/day, with a serum albumin > 30 g/dL, and stable renal function. No response is defined as urinary protein > 3 g/day or a value of 0.6 to 2.9 g/day but serum albumin < 30 g/dL, an increase in serum creatinine ≥ 50 µmol/l or 15% above the base-line value, or the discontinuation of treatment due to side effects.

SECONDARY OUTCOMES:
change in SLEDAI score | 6 months
24-hour urinary protein excretion | 6 months
renal function | 6 months
development of lupus flare (renal or non-renal) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong